CLINICAL TRIAL: NCT02092779
Title: Growth Hormone Deficiency, Empty Sella and Cardio-Metabolic Risk Factors in Obesity: a Cross-Sectional Study.
Brief Title: Growth Hormone Deficiency and Empty Sella Cardio-Metabolic Risk Factors in Obesity: a Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Lucio Gnessi, Associate Professor, University of Roma La Sapienza
Other Study IDs: GHD2014; Dept.Exp.Med.Sapienza.Rome (Other: Sapienza University of Rome)
Record Dates: First submitted 2014-03-17; First posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese patients, no treatment

SUMMARY:
Obesity is a disease not always attributable to nutritional imbalance, frequently associated with changes in key hypothalamic-pituitary (HP) axes. The regain of weight loss after hypochaloric diets has been ascribed to these HP disregulations. The aim of the study is to explore pituitary morphology and its association with pituitary function and metabolic phenotype in outpatient obese individuals evaluated in the period 2010-2013 at the Department of Experimental Medicine of the University of Rome La Sapienza, with features of HP disease in a cross-sectional .

ELIGIBILITY:
Inclusion Criteria:

* Adult obese

Exclusion Criteria:

* psychiatric disturbances, pregnancy, lactation, or drugs known to affect pituitary function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese
Sampling Method: Non-Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2007-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Cranio-caudal pituitary diameter in millimeters | Participants will be followed for the duration of day hospital stay, an expected average of 1 week

SECONDARY OUTCOMES:
Growth hormone releasing hormone plus arginine test for GH secretion μg/L | Participants will be followed for the duration of day hospital stay, an expected average of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Gnessi, MD, PhD, Principal Investigator — University of Roma La Sapienza